CLINICAL TRIAL: NCT02985021
Title: A Phase 2 Study of Docetaxel and Carboplatin for Treatment of Patients With Metastatic, Castration Resistant Prostate Cancer and Germline or Somatic DNA Repair Deficiency
Brief Title: Docetaxel and Carboplatin for Patients With mCRPC and DNA-Repair Deficiencies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Competing studies
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: Prostate Cancer Foundation (Other); VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PugetSoundVA
Record Dates: First submitted 2016-11-22; First posted 2016-12-07 (Estimated); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Hormone-Resistant Prostate Cancer; Metastatic Prostate Carcinoma; Recurrent Prostate Carcinoma; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (docetaxel, carboplatin) (Experimental): Docetaxel 60 mg/m2 will be administered on Day 1 of each 21-day cycle. Carboplatin Area Under the Curve (AUC) 5 will be administered on Day 1 of each 21-day cycle.
  Docetaxel and carboplatin should be administered per institutional guidelines. Treatment will be repeated until disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Docetaxel

INTERVENTIONS:
Drug: Carboplatin — Chemotherapy
  Other Names: Paraplatin
Drug: Docetaxel — Chemotherapy
  Other Names: Taxotere

SUMMARY:
In this study, patients who have metastatic prostate cancer that does not respond to hormone treatment and who have mutations in certain cancer-related genes will be treated with docetaxel and carboplatin chemotherapy.

DETAILED DESCRIPTION:
This is a phase 2 study of the combination of docetaxel and carboplatin in patients with germline inactivation of genes in the homologous recombination pathway, including BRCA1, BRCA2, and Ataxia Telangiectasia Mutated (ATM).

PRIMARY OBJECTIVE To assess rate of 50% Prostate Specific Androgen (PSA) decline to docetaxel and carboplatin

ELIGIBILITY:
Inclusion Criteria

Patients meeting the following inclusion criteria will be eligible to participate in this study:

1. Signed informed consent form (ICF) providing agreement to adhere to the dosing schedule, report for all trial visits and authorization, use and release of health and research trial information.
2. Age > 18 years
3. Known prostate cancer
4. Ongoing gonadal androgen deprivation therapy with gonadotropin-releasing hormone (GnRH) analogues, antagonists or orchiectomy. Patients who have not had an orchiectomy must be maintained on effective GnRH analogue/antagonist therapy.
5. Castration resistant prostate cancer as defined by serum testosterone < 50ng/ml and one of the following:

   * PSA level of at least 2 ng/ml that has risen on at least 2 successive occasions at least 1 week apart.
   * Evaluable disease progression by modified RECIST (Response Evaluation Criteria in Solid Tumors).
   * Progression of metastatic bone disease on bone scan with > 2 new lesions.
6. Prior therapy with abiraterone acetate, enzalutamide, or docetaxel. There is no limit to the number of prior treatment regimens.
7. Presence of metastatic disease on scans.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.
9. Life expectancy >12 weeks.
10. No prior malignancy is allowed except:

    * Adequately treated basal cell or squamous cell skin cancer or
    * In situ carcinoma of any site or
    * Other adequately treated malignancy for which the patient has been disease-free for at least one year (any prior chemotherapy is allowed).
11. Patients must have adequate organ and marrow function as defined below obtained within 14 days prior to start of therapy:

    1. Absolute neutrophil count >1.5 x 109 cells/L
    2. Hgb > 9.0 g/dL
    3. Platelets >100,000 x 109/L
    4. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and total bilirubin levels < 1.5 x Upper Limit of Normal (ULN)
12. Presence of germline inactivation of BRCA1, BRCA2, ATM OR one of the following:

    * Patients with clearly deleterious germline mutations of other genes involved in homologous DNA repair may be included at the investigator's discretion.
    * Patients with homozygous inactivation of genes involved in homologous recombination from primary or metastatic tumor as assessed by a Clinical Laboratory Improvement Amendments (CLIA) level assay for DNA sequencing may be included.
    * Patients with a signature of homologous recombination deficiency in primary or metastatic tissue may be included (VA Puget Sound only).

Exclusion Criteria

Patients who meet any of the following criteria will be excluded from the study:

1. Currently receiving active therapy for other neoplastic disorders.
2. Histologic evidence of small cell carcinoma (morphology alone - immunohistochemical evidence of neuroendocrine differentiation without morphologic evidence is not exclusionary).
3. Prior treatment with platinum-based chemotherapy for prostate cancer.
4. Known parenchymal brain metastasis.
5. Active or symptomatic viral hepatitis or chronic liver disease.
6. Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class II-IV heart disease or cardiac ejection fraction measurement of < 35 % at baseline, if done.
7. Treatment with an investigational therapeutic within 30 days of Cycle 1.
8. Patients with dementia/psychiatric illness/social situations limiting compliance with study requirements or understanding and/or giving of informed consent are not eligible
9. Any medical conditions, which, in the opinion of the investigators, would jeopardize either the patient or the integrity of the data obtained are not eligible.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-11; Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Montgomery, MD, Principal Investigator — VA Puget Sound HCS; Matthew Rettig, MD, Principal Investigator — VA Greater Los Angeles HCS
Locations (3):
- United States (3):
  - VA Greater Los Angeles - West LA, Los Angeles, California
  - VA Ann Arbor Health Care System, Ann Arbor, Michigan
  - VA Puget Sound Health Care System, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Docetaxel, Carboplatin): Docetaxel 60 mg/m2 will be administered on Day 1 of each 21-day cycle. Carboplatin Area Under the Curve (AUC) 5 will be administered on Day 1 of each 21-day cycle.
  Docetaxel and carboplatin should be administered per institutional guidelines. Treatment will be repeated until disease progression or unacceptable toxicity.
  Carboplatin: Chemotherapy
  Docetaxel: Chemotherapy
Period: Overall Study
Arm/Group | Treatment (Docetaxel, Carboplatin)
Started | 2
Completed (Achievement of complete response or 10 cycles of therapy. Patient achieved complete response. One patient did not complete therapy due to inability to comply with study procedures) | 1
Not Completed | 1
Not completed — Inability to comply with study procedures | 1

BASELINE CHARACTERISTICS:
Population: Patients with metastatic, resistant prostate cancer
Arm/Group | Treatment (Docetaxel, Carboplatin)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2
Patients with metastatic resistant prostate cancer [Count of Participants; unit: Participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving >= 50% Reduction in PSA According to Prostate Cancer Working Group 3 (PCWG3) Criteria
Description: Achievement of a PSA50 decline is whether the treatment results in a 50% or greater decline in PSA from baseline PSA prior to therapy
Time Frame: From Day 1 of treatment and up to 30 days after completion of treatment (typically up to 10 cycles of chemotherapy)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Docetaxel, Carboplatin)
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Time Frame: From Day 1 of treatment and up to 30 days after completion of treatment (typically up to 10 cycles of chemotherapy (30 weeks))
Arm/Group | Treatment (Docetaxel, Carboplatin)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT02985021/Prot_SAP_001.pdf
  • Informed Consent Form (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT02985021/ICF_002.pdf